CLINICAL TRIAL: NCT04304235
Title: Smart Triage: Triage and Management of Sepsis in Children Using the Point-of-care Paediatric Rapid Sepsis Trigger (PRST) Tool
Brief Title: Paediatric Rapid Sepsis Trigger (PRST) Tool
Acronym: PRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Kenya Medical Research Institute (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, (John) Ansermino, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: H19-02398
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Sepsis; Infection
Keywords: triage; developing countries
MeSH Terms: conditions — Sepsis; Infections | interventions — Equipment and Supplies; Therapeutics; Guidelines as Topic

STUDY DESIGN:
Intervention Model Description: This is a pre-post intervention study involving pediatric outpatients at Jinja Hospital in Jinja, Uganda, and Mbagathi Hospital in Nairobi, Kenya. The study has three phases: (I) Baseline Period: data is collected on key predictors and outcomes before implementation of the digital triage tool, (II) Interphase Period: model/technology development and usability testing, (III) Intervention Period: data is collected on key predictors and outcomes after implementation of the digital triage tool. Patients who present to the study hospitals in seek of medical care for an acute illness during Phase I will be part of the baseline cohort. Patients who present to the study hospitals in seek of medical care for an acute illness during Phase III will be part of the interventional cohort. A third hospital site, Kiambu Hospital in Nairobi Kenya, will serve as a control hospital, and will only participate in Phase I for the entire duration of the study.
Masking Description: Due to the clinical pre-post intervention design, masking will not be possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Kenya intervention baseline (Active Comparator): Hospital nurses will triage participants using the Emergency Triage and Treatment (ETAT) guidelines, the triage policy that is currently in place at the study hospital sites.
  Interventions: Other: Emergency Triage and Treatment (ETAT) guidelines
- Kenya intervention implementation (Experimental): Hospital nurses will triage participants using the digital triage tool (mhealth intervention).
  Interventions: Device: Pediatric Rapid Sepsis Trigger (PRST) tool
- Kenya control baseline (Active Comparator): Hospital nurses will triage participants using the Emergency Triage and Treatment (ETAT) guidelines, the triage policy that is currently in place at the study hospital sites.
  Interventions: Other: Emergency Triage and Treatment (ETAT) guidelines
- Kenya control implementation (Active Comparator): Hospital nurses will triage participants using the Emergency Triage and Treatment (ETAT) guidelines, the triage policy that is currently in place at the study hospital sites.
  Interventions: Other: Emergency Triage and Treatment (ETAT) guidelines
- Uganda intervention baseline (Active Comparator): Hospital nurses will triage participants using the Emergency Triage and Treatment (ETAT) guidelines, the triage policy that is currently in place at the study hospital sites.
  Interventions: Other: Emergency Triage and Treatment (ETAT) guidelines
- Uganda intervention implementation (Experimental): Hospital nurses will triage participants using the digital triage tool (mhealth intervention)
  Interventions: Device: Pediatric Rapid Sepsis Trigger (PRST) tool
- Uganda control implementation (Active Comparator): Hospital nurses will triage participants using the Emergency Triage and Treatment (ETAT) guidelines, the triage policy that is currently in place at the study hospital sites.
  Interventions: Other: Emergency Triage and Treatment (ETAT) guidelines

INTERVENTIONS:
Device: Pediatric Rapid Sepsis Trigger (PRST) tool — The digital platform consists of a mobile application integrating a pulse oximetry sensor attached to this device, with embedded smart algorithms that predict a critically ill state, or level of risk (below) in a child presenting at the hospital. The platform also includes an interactive dashboard located in strategic locations (e.g., laboratory, consultation rooms), which connects to the mobile application through a secure local network and displays the triage data to provide real-time monitoring for the physicians who manage the patients.
  Arms: Kenya intervention implementation; Uganda intervention implementation
Other: Emergency Triage and Treatment (ETAT) guidelines — These are the triage guidelines currently applied in the study hospital sites. This will be the comparator group.
  Arms: Kenya control baseline; Kenya control implementation; Kenya intervention baseline; Uganda control implementation; Uganda intervention baseline

SUMMARY:
Sepsis is the leading cause of death and disability in children, every hour of delay in treatment is associated with greater organ damage and ultimately death. The challenges, especially in poor countries, are the delays in diagnosis and the inability to identify children in urgent need of treatment.To circumvent these challenges, we propose the development and clinical evaluation of a trigger tool that will reduce the time to diagnosis and prompt the timely initiation of life-saving treatment. The key innovations are 1) a data-driven approach to rapid diagnosis of sepsis severity and 2) a low- cost digital tagging system to track the time to treatment. The tool will require minimal cost, clinical expertise and training or time to use.

The tool will identify high risk children and reduce time to treatment. The digital platform (mobile device and dashboard) will create a low-cost, highly scalable solution for children with sepsis.

DETAILED DESCRIPTION:
This is a pre-post intervention study involving pediatric patients presenting to the study hospitals in seek of medical care for an acute illness. The study involves three phases: (I) Baseline Period, (II) Interphase Period, (III) Intervention Period.

Phase I (3-6 months) will be a prospective observational cohort at Mbagathi County Hospital in Nairobi, Kenya, and Jinja Regional Referral Hospital in Jinja, Uganda. During this period, there will be no changes to healthcare delivery procedures in the study hospitals. Triage will continue to be performed by hospital staff using Emergency Triage and Treatment (ETAT) guidelines, the system that is currently in effect at the study hospitals. Data collection will be undertaken in the triage waiting area. While participants are waiting for their turn to be seen by the hospital triage nurses, our trained study nurses will collect data on a pre-selected list of predictor variables. These data will be used to develop a clinical prediction model based on the need for hospital admission.

Control Site (Phase I, 12 months): Kiambu County Referral Hospital in Nairobi, Kenya will serve as the control site and no intervention will be implemented. At this site, Phase I will commence for a period of 12 months. There will be no Phase II or Phase III.

Phase II (1-3 months) will involve technology development, usability testing, and training.

Phase IIa: Technology Development. A risk prediction model will be derived using the data collected in Phase I and implemented in a Digital Triaging Platform, along with a digitized version of the ETAT+ guidelines. The Digital Triaging Platform, including vital sign measurement devices (PhoneOx and RRate and the mobile application and clinical dashboard has already been developed and evaluated. Once the digital triage tool has been developed, it will be evaluated in potential users using simulated patient scenarios and a 'Think Aloud' method.

Phase IIb: Usability Testing and Training. The digital triage tool will be evaluated for ease of interface navigation, functionality and basic workflow. A sample of 15 health workers in the study hospitals to represent the primary user groups will be selected for participation in the 60-minute-long usability testing initiatives. Participants will be recruited through word of mouth as there is a very small cadre of potential participants. The objective of the training is to (1) ensure healthcare workers understand how to correctly collect and interpret patient information, and (2) to obtain feedback on the digitization of the tool. Training will use a framework that meets key international norms for testing digital tools, including, the think-aloud method and a questionnaire.

Each training session will be conducted by a moderator and observer. During the evaluation, the observer will be seated next to the participant and will record user interaction with each interface, comments, errors, and duration of each task. Participants will be given 3-5 patient scenarios which will list hypothetical information to be entered into the app. This information will be designed to represent routine data collected during triage examination at the study hospitals. The moderator will provide the fictional charts to participants and instruct them throughout the tasks. During the simulated patient scenarios, participants will be asked to think aloud, in order to assess their thought process as they used the app. Participants will be specifically instructed to comment on the layout of the app screen, the dialogue on each interface, the order of tasks, and any additional observations or opinions. After learning the basics of the digital platform, the participants will be read the think aloud instructions and asked to perform the list of tasks and answer questions. The observer will complete a checklist to ensure that all tasks were completed, questions will be asked to evaluate task comprehension, and notes will be taken about whether help was needed in completing each task. At the end of the training session, participants will complete a triage tool training questionnaire to provide an understanding of the practical benefits and drawbacks of incorporating the digital triage tool into a clinical context. The questionnaire will utilize open ended questions and comment responses. from this evaluation. Responses from the survey will be anonymous. The data generated from the training phase is fictitious and will not be linked to any individual subject.

Transcriptions and Think Aloud observations will be analyzed using the Framework Method to assess attitudes of health workers. Responses will be transcribed and coded for the identification, examination and interpretation of emerging themes and patterns. Results from the analysis, feedback from the questionnaires, and comments on the observer checklists will be used to generate a report with suggested improvements to be shared with the quality improvement implementation team prior to Phase III.

Phase III (3-6 months) will be an interventional period involving routine use of the digital triage tool by the hospital triage nurses at Mbagathi County Hospital in Nairobi, Kenya, and Jinja Regional Referral Hospital in Jinja, Uganda. The digital triage tool will not replace triage policies already in place at the study hospitals, but rather it will supplement and strengthen existing triage systems. As done in Phase I, study nurses will collect data on the pre-selected list of predictor variables in the triage waiting area while participants are waiting to be seen by the hospital triage nurses (who will be using the digital triage tool). Continued collection of predictor variables will allow comparison of participant characteristics in the pre-intervention cohort and the post-intervention cohort. (Funder: Wellcome Trust Innovator Award # 215695/Z/19/Z)

ELIGIBILITY:
Inclusion Criteria:

* All paediatric outpatients presenting to the study hospitals for medical treatment. The lower age limit will include children aged from 0 days, and the upper age limit will be in accordance to respective hospitals' practice for paediatric admissions (this may be 12, 15 or 19 years).
* Informed parental/guardian consent provided.
* Assent from children older than 13 years in addition to parental/guardian consent provided.

Exclusion Criteria:

-Patients presenting to the outpatient department for elective cases (e.g. elective surgery or change of dressing) or for clinical review appointment.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18693 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Ansermino, Principal Investigator — The University of British Columbia
Locations (3):
- Kenya (2):
  - Kiambu County Referral Hospital, Nairobi
  - Mbagathi County Hospital, Nairobi
- Jinja Regional Referral Hospital, Jinja, Uganda

IPD SHARING:
Plan to Share IPD: Yes
After the study period, a de-identified copy of the data will be prepared for deposition in a repository with open access with proper governance mechanisms. We will make every effort to prevent re-identification of subjects by coding data that has the potential of being identifiable. The de-identified study data will be made publicly available using the Harvard Dataverse (https://dataverse.harvard.edu/), which is the data repository for KWTRP, and a URL will be made accessible. To enhance visibility, sharing and collating datasets with other collaborating sites for increased usability/re-use, de-identified will also be shared availed to reputable data hosting service such as the INDEPTH Data Repository (http://www.indepth-ishare.org/index.php/home), or through the newly established Pediatric Sepsis CoLab (sponsored by the World Federation of Pediatric Critical and Intensive care Societies).
Time Frame: Data will be made available within 12 months following completion of the study.
Access Criteria: Sharing and access will be managed and subject to institutional agreements (Kenya Medical Research Institute, The University of British Columbia, Makerere University School of Public Health) that will set terms for how requests and access will be managed. We will ensure that a rigorous data governance structure is used by the data hosting service. The distribution will only occur with agreement from Principal Investigators and the investigators at all of the study sites.

REFERENCES:
- [Result] Ansermino JM, Pillay Y, Tagoola A, Zhang C, Dunsmuir D, Kamau S, Kigo J, Agaba C, Aye IA, Hwang B, Novakowski SK, Huxford C, Wiens MO, Kimutai D, Ouma M, Ahmed I, Mwaniki P, Oyella F, Tenywa E, Nambuya H, Toliva BO, Kenya-Mugisha N, Kissoon N, Akech S; Pediatric Sepsis CoLab. Implementation of Smart Triage combined with a quality improvement program for children presenting to facilities in Kenya and Uganda: An interrupted time series analysis. PLOS Digit Health. 2025 Mar 10;4(3):e0000466. doi: 10.1371/journal.pdig.0000466. eCollection 2025 Mar. PMID 40063663
- [Derived] Li ECK, Tagoola A, Komugisha C, Nabweteme AM, Pillay Y, Ansermino JM, Khowaja AR. Cost-effectiveness analysis of Smart Triage, a data-driven pediatric sepsis triage platform in Eastern Uganda. BMC Health Serv Res. 2023 Aug 31;23(1):932. doi: 10.1186/s12913-023-09977-5. PMID 37653477
- [Derived] Li ECK, Grays S, Tagoola A, Komugisha C, Nabweteme AM, Ansermino JM, Mitton C, Kissoon N, Khowaja AR. Cost-effectiveness analysis protocol of the Smart Triage program: A point-of-care digital triage platform for pediatric sepsis in Eastern Uganda. PLoS One. 2021 Nov 17;16(11):e0260044. doi: 10.1371/journal.pone.0260044. eCollection 2021. PMID 34788338
- [Derived] Mawji A, Li E, Komugisha C, Akech S, Dunsmuir D, Wiens MO, Kissoon N, Kenya-Mugisha N, Tagoola A, Kimutai D, Bone JN, Dumont G, Ansermino JM. Smart triage: triage and management of sepsis in children using the point-of-care Pediatric Rapid Sepsis Trigger (PRST) tool. BMC Health Serv Res. 2020 Jun 3;20(1):493. doi: 10.1186/s12913-020-05344-w. PMID 32493319
- Available data/document: Individual Participant Data Set: doi.org/10.5683/SP3/SIL — https://borealisdata.ca/dataverse/smart_triage — Open access to all study materials and data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at hospitals in two countries . Each country had a control and intervention site. A baseline period of data collection occurred at all sites except the control site in Uganda (due to COVID 19 pandemic restrictions).
  Kenya: Intervention site Baseline, Kenya Intervention site Implementation, Kenya Control site Baseline, Kenya Control site Implementation
  Uganda: Intervention site Baseline, Uganda Intervention site Implementation, Uganda Control site Implementation:
Pre-assignment Details: Non infectious illness, routine clinic visit
Period: Overall Study
Arm/Group | Kenya Intervention Baseline | Kenya Intervention Implementation | Kenya Control Baseline | Kenya Control Implementation | Uganda Intervention Baseline | Uganda Intervention Implementation | Uganda Control Implementation
Started (Baseline) | 2856 | 3497 | 2520 | 3177 | 1697 | 2026 | 2920
Completed | 2856 | 3428 | 2520 | 3177 | 1408 | 1903 | 2855
Not Completed | 0 | 69 | 0 | 0 | 289 | 123 | 65
Not completed — incomplete triage data | 0 | 69 | 0 | 0 | 289 | 123 | 65

BASELINE CHARACTERISTICS:
Population: same as Participant Flow information
Groups:
- Kenya Intervention Baseline: Baseline cohort at Kenya intervention site
- Kenya Intervention Implementation: Implementation cohort at Kenya implementation site
- Kenya Control Baseline: Baseline cohort at Kenya control site
- Kenya Control Implementation: Implementation cohort at Kenya control site
- Uganda Intervention Baseline: Baseline cohort at Uganda intervention site
- Uganda Intervention Implementation: Implementation cohort at Uganda implementation site
- Uganda Control Implementation: Implementation cohort at Uganda control site
- Total: Total of all reporting groups
Arm/Group | Kenya Intervention Baseline | Kenya Intervention Implementation | Kenya Control Baseline | Kenya Control Implementation | Uganda Intervention Baseline | Uganda Intervention Implementation | Uganda Control Implementation | Total
Number analyzed (Participants) | 2856 | 3428 | 2520 | 3177 | 1408 | 1903 | 2855 | 18147
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 25 [10.3 to 54.7] | 31.2 [11 to 62.2] | 17.55 [7.85 to 32.8] | 13.3 [5.8 to 30.2] | 13.55 [6.5 to 31] | 15 [7.3 to 30.3] | 17.3 [7.9 to 39.2] | 22.4 [7.2 to 47.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1252 | 1466 | 1207 | 1504 | 676 | 908 | 1418 | 8431
  Male | 1604 | 1962 | 1313 | 1673 | 732 | 995 | 1437 | 9716
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Time to antimicrobial administration [Median (Inter-Quartile Range); unit: Minutes] — This study is not a randomized trial. Each cohort has bassline observations however the time to antibiotic administration is an outcome. This is reported as an outcome
  Minutes | 115 [68 to 203] | 123 [68 to 213] | 239 [160 to 388] | 261 [193 to 392] | 255 [186 to 348] | 239 [171 to 303] | 212 [129 to 295] | 206 [114 to 298]

OUTCOME MEASURES:

1. Primary Outcome: Time to Administration of an Appropriate Antimicrobial
Description: Time in minutes to administer an appropriate antimicrobial, which includes at least one antibiotic or antimalarial (treatment determined and administered by hospital staff). The time is measured from when the child arrives at the facility (time of the first registration) until the antimicrobial administration is started.
Time Frame: 1 day
Population: Children presenting to the outpatient department at facility
Measure: Mean (Inter-Quartile Range); unit: minutes
Groups:
- Kenya Intervention Implementation: Implementation cohort at the Kenya intervention site
- Kenya Control Baseline: Baseline cohort at the Kenya control site
- Kenya Control Implementation: Implementation cohort at the Kenya control site
- Uganda Intervention Implementation: Implementation cohort at the Uganda intervention site
Arm/Group | Kenya Intervention Baseline | Kenya Intervention Implementation | Kenya Control Baseline | Kenya Control Implementation | Uganda Intervention Baseline | Uganda Intervention Implementation | Uganda Control Implementation
Number analyzed (Participants) | 2856 | 3428 | 2520 | 3177 | 1408 | 1903 | 2855
minutes | 115 [68 to 203] | 123 [68 to 213] | 239 [160 to 388] | 261 [193 to 392] | 255 [186 to 348] | 239 [171 to 303] | 212 [129 to 295]

2. Other Pre Specified Outcome: Readmission
Description: The child is readmitted to the hospital after being discharged
Time Frame: 7 days
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Sites: Number of readmissions at baseline sites
- Control Sites: Number of readmissions at control sites
- Intervention Sites: Number of admissions at intervention sites
Arm/Group | Baseline Sites | Control Sites | Intervention Sites
Number analyzed (Participants) | 4264 | 8552 | 5331
Participants | 57 | 57 | 48

3. Other Pre Specified Outcome: Mortality
Description: Death within 7 days
Time Frame: 7 days
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Sites: Number of deaths at baseline sites
- Control Sites: Number of deaths at control sites
- Intervention Sites: Number of deaths at intervention sites
Arm/Group | Baseline Sites | Control Sites | Intervention Sites
Number analyzed (Participants) | 4264 | 8552 | 5331
Participants | 39 | 23 | 14

4. Other Pre Specified Outcome: Admission
Description: Admission to hospital
Time Frame: 12 hours
Population: All enrolled children
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Sites: Number of admissions at baseline sites
- Control Sites: Number of admissions at control sites
Arm/Group | Baseline Sites | Control Sites | Intervention Sites
Number analyzed (Participants) | 4264 | 8552 | 5331
Participants | 581 | 474 | 452
Statistical Analysis 1: Comparison: Baseline Sites vs Control Sites vs Intervention Sites; Test type: Superiority; Odds Ratio (OR) = 2.22

5. Other Pre Specified Outcome: Clinical Diagnosis
Description: The clinical diagnosis for each participant
Time Frame: 12 hours
Population: All participants.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Sites: Number of diagnoses at bassline
- Control Sites: Number of diagnoses at control sites
- Intervention Sites: Number of diagnoses at intervention sites
Arm/Group | Baseline Sites | Control Sites | Intervention Sites
Number analyzed (Participants) | 567 | 472 | 451
Participants
  Malaria | 131 | 100 | 85
  Pneumonia | 139 | 154 | 104
  Broncholitis | 3 | 5 | 2
  Diarrhea/ Gastro | 15 | 12 | 12
  Meningitis | 11 | 6 | 5
  Malnutrition | 17 | 5 | 8
  Septicemia | 58 | 23 | 75
  Neonatal sepsis | 12 | 32 | 17
  Dehydration | 20 | 12 | 20
  Other | 161 | 123 | 123

6. Other Pre Specified Outcome: Length of Stay
Description: Length of stay in hospital for admitted cases
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Baseline Sites; Control Sites; Intervention Sites: Length of stay in days
Arm/Group | Baseline Sites | Control Sites | Intervention Sites
Number analyzed (Participants) | 581 | 474 | 452
Days | 4 [2 to 7] | 4 [3 to 6] | 4 [2 to 6]

7. Post Hoc Outcome: Number of Intravenous Antimicrobials in Admitted Cases
Description: Number cases receiving antimicrobials in the cohort of admitted cases
Time Frame: 24 hours
Population: Participants admitted to hospital
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Sites; Control Sites; Intervention Sites: Number of cases receiving antimicrobials
Arm/Group | Baseline Sites | Control Sites | Intervention Sites
Number analyzed (Participants) | 581 | 474 | 452
Participants | 512 | 361 | 406

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Kenya Intervention Implementation: Implementation cohort at Kenya intervention site
- Uganda Intervention Implementation: Implementation cohort at Uganda intervention site
Arm/Group | Kenya Intervention Baseline | Kenya Intervention Implementation | Kenya Control Baseline | Kenya Control Implementation | Uganda Intervention Baseline | Uganda Intervention Implementation | Uganda Control Implementation
All-Cause Mortality (participants affected / at risk) | 29/2856 | 10/3428 | 11/2520 | 10/3177 | 11/1408 | 4/1903 | 2/2855
Serious Adverse Events (participants affected / at risk) | 0/2856 | 0/3428 | 0/2520 | 0/3177 | 0/1408 | 0/1903 | 0/2855
Other Adverse Events (participants affected / at risk) | 0/2856 | 0/3428 | 0/2520 | 0/3177 | 0/1408 | 0/1903 | 0/2855

LIMITATIONS AND CAVEATS:
Simultaneous recruitment across countries disrupted by COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04304235/Prot_SAP_ICF_000.pdf